CLINICAL TRIAL: NCT00002641
Title: RANDOMISED TRIAL OF ADJUVANT CHEMOTHERAPY WITH HIGH-DOSE DOXORUBICIN, IFOSFAMIDE AND LENOGRASTIM IN HIGH GRADE SOFT TISSUE SARCOMA
Brief Title: Surgery With or Without Chemotherapy in Treating Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-62931; EORTC-62931; CAN-NCIC-SR3
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2002-07

CONDITIONS: Endometrial Cancer; Kidney Cancer; Ovarian Cancer; Pheochromocytoma; Sarcoma
Keywords: adult angiosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult neurofibrosarcoma; adult synovial sarcoma; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; adult alveolar soft-part sarcoma; adult epithelioid sarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; adult malignant mesenchymoma; adult rhabdomyosarcoma; localized benign pheochromocytoma; regional pheochromocytoma; recurrent pheochromocytoma; stage II uterine sarcoma; stage III uterine sarcoma; recurrent uterine sarcoma; uterine carcinosarcoma; uterine leiomyosarcoma; endometrial stromal sarcoma; ovarian sarcoma; clear cell sarcoma of the kidney; stage II adult soft tissue sarcoma
MeSH Terms: conditions — Endometrial Neoplasms; Kidney Neoplasms; Ovarian Neoplasms; Pheochromocytoma; Sarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Sarcoma, Synovial; Sarcoma, Alveolar Soft Part; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Malignant mesenchymal tumor; Rhabdomyosarcoma; Sarcoma, Endometrial Stromal | interventions — Filgrastim; Doxorubicin; Ifosfamide; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: doxorubicin hydrochloride
Drug: ifosfamide
Drug: isolated perfusion
Procedure: adjuvant therapy
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether giving chemotherapy after surgery is more effective than surgery alone in treating soft tissue sarcoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery with or without chemotherapy in treating patients who have soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the local disease control, overall survival, and relapse-free survival in patients with high-grade soft tissue sarcoma treated with adjuvant high-dose doxorubicin and ifosfamide plus filgrastim (G-CSF) vs no adjuvant chemotherapy and G-CSF after definitive surgery.
* Compare the toxicity and morbidity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, site of primary tumor (extremity vs trunk, including shoulder, pelvic girdle, head, or neck vs central, including intrathoracic, visceral, uterine, or retroperitoneal), size of primary tumor (less than 5 cm vs 5 cm or greater in largest diameter), postoperative radiotherapy (yes vs no), and isolated limb perfusion therapy (yes vs no).

Some patients undergo isolated limb perfusion therapy with cytotoxics and/or cytokines.

No more than 8 weeks after biopsy or inadequate surgery, patients undergo definitive surgery. Patients with complete resection undergo radiotherapy assessment and then randomization. Patients with incomplete or marginal resection (except for central lesions) undergo re-excision and, in the absence of macroscopic disease, assessment for postoperative radiotherapy followed by randomization.

* Randomization: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive no adjuvant chemotherapy or filgrastim (G-CSF). Beginning within 6 weeks after surgery, eligible patients undergo radiotherapy as outlined below.
  * Arm II: Beginning within 4 weeks after surgery, patients receive high-dose doxorubicin IV over 20 minutes followed by ifosfamide IV over 24 hours and G-CSF subcutaneously daily beginning 24 hours after completion of ifosfamide infusion and continuing for 10 days. Treatment continues every 3 weeks for 5 courses. Beginning within 6 weeks after completion of chemotherapy, eligible patients undergo radiotherapy as outlined below.
* Radiotherapy: Patients with incomplete or marginal resection undergo radiotherapy 5 days a week for 6-6.6 weeks. Patients with complete microscopic resection undergo radiotherapy 5 days a week for 5 weeks followed by boost radiotherapy 5 days a week for 1 week.

Patients are followed every 2 months for 1 year, every 3 months for 2 years, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 350 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven soft tissue sarcoma that is amenable to definitive surgery no more than 8 weeks after biopsy or inadequate surgery

  * Eligible subtypes:

    * Alveolar soft part sarcoma
    * Angiosarcoma
    * Fibrosarcoma
    * Leiomyosarcoma
    * Malignant fibrous histiocytoma
    * Liposarcoma (round cell and pleomorphic)
    * Miscellaneous sarcoma (including pelvic mixed mesodermal tumors)
    * Malignant paraganglioma
    * Neurogenic sarcoma
    * Rhabdomyosarcoma
    * Synovial sarcoma
    * Unclassifiable sarcoma
  * Ineligible subtypes:

    * Chondrosarcoma
    * Dermatofibrosarcoma
    * Embryonal rhabdomyosarcoma
    * Ewing's sarcoma
    * Kaposi's sarcoma
    * Liposarcoma (myxoid and well differentiated)
    * Malignant mesothelioma
    * Neuroblastoma
    * Osteosarcoma
* Confirmed high-grade tumor (i.e., Trojani Grade II or III)
* No metastases on staging with chest x-ray and thoracic CT scan
* No regional lymph node involvement
* Locally recurrent disease allowed

  * Interval of 3 months or more between definitive surgery and recurrence

PATIENT CHARACTERISTICS:

Age:

* 16 to 69

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm^3
* Platelet count greater than 120,000/mm^3
* No bleeding disorders

Hepatic:

* Bilirubin no greater than 1.25 times normal
* No severe hepatic dysfunction

Renal:

* Creatinine less than 1.6 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No clear history of angina
* No documented myocardial infarction
* No existing cardiac failure

Other:

* No serious infection
* No other malignancy except adequately treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior systemic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to affected area

Surgery:

* See Disease Characteristics

Ages: 16 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 1995-02; Primary Completion 2006-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Penella J. Woll, MD, PhD, Study Chair — Cancer Research Centre at Weston Park Hospital; Vivien H.C. Bramwell, MB, BS, PhD, FRCP, Study Chair — Tom Baker Cancer Centre - Calgary
Locations (45):
- Karl-Franzens-University Graz, Graz, Austria
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Canada (11):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University, Montreal, Quebec
- Denmark (2):
  - Aarhus Kommunehospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (3):
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - Institut Gustave Roussy, Villejuif
- Germany (5):
  - Robert Roessle Klinik, Berlin
  - Universitaetsklinikum Essen, Essen
  - Universitaets-Krankenhaus Eppendorf, Hamburg
  - Klinikum Grosshadern, Munich
  - Eberhard Karls Universitaet, Tübingen
- Istituto Nazionale per lo Studio e la Cura dei Tumori, Milano (Milan), Italy
- Netherlands (3):
  - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - Daniel Den Hoed Cancer Center at Erasmus University Medical Center, Rotterdam
- Instituto Portugues de Oncologia de Francisco Gentil - Centro de Lisboa, Lisbon, Portugal
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Hospital de la Santa Cruz I Sant Pau, Barcelona, Spain
- Switzerland (3):
  - Inselspital, Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - St. Gallen, Sankt Gallen
- United Kingdom (8):
  - Royal Devon and Exeter Hospital, Exeter, England
  - St. James's Hospital, Leeds, England
  - Royal Marsden NHS Trust - London, London, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Weston Park Hospital, Sheffield, England

REFERENCES:
- [Background] Le Cesne A, Van Glabbeke M, Woll PJ, et al.: The end of adjuvant chemotherapy (adCT) era with doxorubicin-based regimen in resected high-grade soft tissue sarcoma (STS): pooled analysis of the two STBSG-EORTC phase III clinical trials. [Abstract] J Clin Oncol 26 (Suppl 15): A-10525, 2008.
- [Derived] Woll PJ, Reichardt P, Le Cesne A, Bonvalot S, Azzarelli A, Hoekstra HJ, Leahy M, Van Coevorden F, Verweij J, Hogendoorn PC, Ouali M, Marreaud S, Bramwell VH, Hohenberger P; EORTC Soft Tissue and Bone Sarcoma Group and the NCIC Clinical Trials Group Sarcoma Disease Site Committee. Adjuvant chemotherapy with doxorubicin, ifosfamide, and lenograstim for resected soft-tissue sarcoma (EORTC 62931): a multicentre randomised controlled trial. Lancet Oncol. 2012 Oct;13(10):1045-54. doi: 10.1016/S1470-2045(12)70346-7. Epub 2012 Sep 4. PMID 22954508